CLINICAL TRIAL: NCT05963906
Title: An Innovative, Accessible, and Flexible Approach for Household Food Waste Measurement - SCFI
Brief Title: Food Survey, Curbside, Remote APPs SCFI
Acronym: FoodSCRAPPSCFI
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Martin, Corby, K., M.D. (Individual)
Responsible Party: Principal Investigator, John Apolzan, Associate Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-007 B
Record Dates: First submitted 2023-07-14; First posted 2023-07-27 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Nutrition Sciences; Climate; Recycling; Waste Management

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SCFI: SCFI participants will complete a survey once per week for three consecutive weeks. They will participate in training for the FoodImage app and deploy it the last two weeks of their study period. During these last two weeks, these participants will also have waste collected on designated days by a waste pickup contractor.

SUMMARY:
The proposed research will create accurate and standardized household food waste measurement technologies that foster serial and longitudinal assessments as well as confident and convenient one-time measurement. The investigators propose the SCFI field study where participants simultaneously deploy 3 measurement approaches (1) retrospective surveys (2) curbside audits, and (3) the FoodImage smartphone app.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, age 18-64 years
* Willing and able to store household food waste for curbside pickup by a third-party waste pickup company
* Internet or Wi-Fi availability to complete online surveys
* Ownership of an IPhone 9s or later, operable Apple ID, password, and email address that they are willing and able to use to collect data during the study. Subject acknowledges data usage and associated charges are a result of study
* Willing to complete all study procedures and adhere to study visit timelines

Exclusion Criteria:

* Not willing to adhere to study procedures and study visit timelines
* Any condition or circumstance that in the judgement of the PI could interfere with study participation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be from the greater Columbus, OH and Baton Rouge, LA areas.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Household Food Waste | 1 week
  Weight
Household Food Waste | 1 week
  Energy (kcal)

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (2):
- United States (2):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication after a DTA with the institution. Please provide a research question.
Supporting Information: Study Protocol, ICF